CLINICAL TRIAL: NCT01069952
Title: Electrical Stimulation of the Internal Capsule for Intractable Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Dr. Benjamin Greenberg, Chief of Outpatient Services, Associate Professor of Psychiatry, Butler Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G010351; 0201-001 (Other: Butler Hospital IRB)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Depression
Keywords: Deep Brain Stimulation; Treatment Refractory; Neurosurgery; Implantable Neurostimulator (INS); Internal Capsule
MeSH Terms: conditions — Depression | interventions — Implantable Neurostimulators

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active DBS (Experimental): Participants will receive deep brain stimulation.
  Interventions: Device: Deep Brain Stimulation System

INTERVENTIONS:
Device: Deep Brain Stimulation System — In DBS, thin wires are used to carry electric current to the parts of the brain involved in depression symptoms. These wires are implanted surgically and are attached to battery operated stimulators usually implanted in the chest. The study doctor will adjust the settings of the electrical stimulation to optimize treatment for each participant.
  Other Names: Deep Brain Stimulation System from Medtronic, Inc.; Implantable Neurostimulator (INS)

SUMMARY:
This study will evaluate the safety and efficacy of deep brain stimulation in treating people with several and otherwise treatment-resistant depression.

DETAILED DESCRIPTION:
Despite the availability of effective treatments, a substantial portion of patients fail to recover from episodes of depression. Assuming a conservative rate of 20%, and given the prevalence of major depression in the general population, over 3.5 million Americans would be expected to manifest refractory illness if all those with depression received treatment. Although rarely used in the U.S., neurosurgical approaches to severely refractory depression have shown efficacy in a number of uncontrolled studies, primarily from European investigators. Deep brain stimulation (DBS) is a procedure that involves the use of thin wires to carry electric current to parts of the brain associated with producing depression symptoms. DBS has been effectively and safely used to treat movement disorders, such as Parkinson's disease, and may be beneficial in reducing depression symptom severity. This study will evaluate the safety and efficacy of DBS in treating people with severe and treatment-resistant depression.

Study participation through follow-up will last up to three years. Participants will be allowed to remain on any pre-surgical medications or behavioral therapy programs throughout the study. Before surgery, all participants will undergo a series of initial tests and examinations that will include a physical and neurological examination; laboratory testing to screen for significant hematologic, hepatic, renal or endocrine abnormalities; and detailed psychological testing including tests of perception, learning, and memory.

Implantation of all devices will be preformed at a single session. The patient will undergo local anesthesia for the implantation of the leads, and the implanted pulse generator will be implanted under general anesthesia. On the day of the surgery, participants will have a metal frame fixed to their heads for support during surgery. Using coordinates individually determined by preoperative MRI, a pair of tetrapolar leads will be inserted into the anterior limb of each internal capsule and fixed to the skull with a burr hole ring and cap. The leads will be inserted so that the stimulation sites span the dorsal-ventral extent of the anterior capsule or target the ventral half of the anterior capsule.

After placement of the DBS system, the patient will be admitted to the hospital for overnight evaluation for possible complications of the procedure, including possible hemorrhage or infection. Postoperative evaluation will consist of physical and neurological examinations, postoperative CBC, electrolyte panel, plain x-ray studies of head, neck, and chest including a standard shunt series to ensure integrity of connections and to document positioning of stimulating hardware. A head CT scan will be obtained within 24 hours postoperatively to monitor for possible postoperative intracranial hemorrhage.

If none of the above complications occur, the patient will be discharged home the following day with the DBS system off to allow resolution of the cellular reactions to electrode placement. Three weeks after placement of the DBS system, the patient will return to being the outpatient phase of testing the effects of stimulation.

During the intensive outpatient phase of the study, each of the outpatient visits will last approximately two hours. These are anticipated to occur at from 1 to 5 day intervals. On each day, we will do a brief clinical interview and obtain structured ratings of depressive symptoms, mood and affect, possible side effects, and cognition.

After completion of the two year study, patients will be given the choice of continued DBS, for a total of three years after implantation, or until the stimulator batteries fail. Patients will also be offered alternative treatment, outside of this study, including anterior capsulotomy, depending on availability given the patient's financial circumstances and insurance coverage, or further conventional therapy. Long-term patient follow-up will continue indefinitely where possible.

During this study, patients will also be invited to undergo a series of three Positron Emission Tomography (PET) scans under a separate IRB protocol at Massachusetts General Hospital, to assess the effects of capsular stimulation on activity in brain circuits implicated in depression. Subjects' participation in this separate protocol is not a condition for entering the DBS study.

ELIGIBILITY:
Inclusion Criteria:

* Major depression, severe, unipolar type, diagnosed by Structural Clinical Interview for DSM-IV (SCID-IV), judged to be of disabling severity.
* 24-item Hamilton Depression Rating Scale (HDRS) of at least 21.
* Global Assessment of Function (GAF) score of 45 or less.
* A recurrent (greater than or equal to 4 episodes) or chronic (episode duration greater than or equal to two years) course and a minimum of 5 years since the onset of the first depressive episode. Major impairment in functioning or potentially severe medical outcomes (repeated hospitalizations, serious suicidal or other self-injurious behavior).
* Failure to respond to respond to:

  1. Adequate trials (greater than or equal to 6 weeks at the maximum recommended or tolerated dose) of primary antidepressants from at least 3 different classes and;
  2. Adequate trials (greater than or equal to 4 weeks at the usually recommended or maximum tolerated dose of augmentation/combination of a primary antidepressant using at least 2 different augmenting/combination agents (lithium, T3, stimulants, neuroleptics, anticonvulsants, buspirone, or a second primary antidepressant) and;
  3. An adequate trial of individual psychotherapy (greater than or equal to 20 sessions with an experienced psychotherapist)
* Age 18 to 65 years
* Able to comply with the operational and administrative requirements of participation in the study.
* Able to give written informed consent.
* Either drug-free or on a stable drug regimen for at least 6 weeks at the time of entry into the study.
* Good general health.

Exclusion Criteria:

* Current or past non-affective psychotic disorder.
* Any current clinically significant neurological disorder or medical illness affecting brain function, other than motor tics or Gilles de la Tourette syndrome.
* Any clinically significant abnormality on preoperative magnetic resonance imaging (MRI).
* Any surgical contraindications to undergoing DBS, including labeled contraindications for DBS and/or inability to undergo pre-surgical MRI (cardiac pacemaker, pregnancy, metal in body, severe claustrophobia), infection coagulopathy, inability to undergo an awake operation, significant cardiac or other medical risk factors for surgery.
* Current or unstably remitted substance abuse.
* Pregnancy and women of childbearing age not using effective contraception.
* History of severe personality disorder.
* Imminent risk of suicide (based on the judgment of the investigators).
* Not able to comply with the operational and administrative requirements of participation in the study (based on the judgment of the investigators).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2002-12; Primary Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | Administered at base line, every 1 to 5 days during the acute phase (2 months), monthly during the chronic phase, then every three months during the open continuation phase

SECONDARY OUTCOMES:
Inventory for Depressive Symptoms, Self Report (IDS-SR) | Administered at base line, every 1 to 5 days during the acute phase (2 months), monthly during the chronic phase, then every three months during the open continuation phase

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Greenberg, MD, PhD, Principal Investigator — Butler Hospital/Brown University
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Result] Malone DA Jr, Dougherty DD, Rezai AR, Carpenter LL, Friehs GM, Eskandar EN, Rauch SL, Rasmussen SA, Machado AG, Kubu CS, Tyrka AR, Price LH, Stypulkowski PH, Giftakis JE, Rise MT, Malloy PF, Salloway SP, Greenberg BD. Deep brain stimulation of the ventral capsule/ventral striatum for treatment-resistant depression. Biol Psychiatry. 2009 Feb 15;65(4):267-75. doi: 10.1016/j.biopsych.2008.08.029. Epub 2008 Oct 8. PMID 18842257
- [Result] Carpenter LL, Friehs GM, Tyrka AR, Rasmussen S, Price LH, Greenberg BD. Vagus nerve stimulation and deep brain stimulation for treatment resistant depression. Med Health R I. 2006 Apr;89(4):137, 140-1. PMID 16676910